CLINICAL TRIAL: NCT05793866
Title: The Effect of Buteyko Breathing Technique on Asthma Control and Quality of Life in Children Aged 7-12 With Asthma
Brief Title: The Effect of Buteyko Breathing Technique on Asthma Control and Quality of Life in Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Emel Yürük, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BALCALI HOSPITAL
Record Dates: First submitted 2023-02-03; First posted 2023-03-31 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Asthma in Children
Keywords: Asthma; Quality of Life; Asthma Control
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUTEYKO RESPIRATORY TECHNIQUE APPLIED GROUP (Experimental): This group consists of children between the ages of 7 and 12 who are being treated for asthma. Children with written and verbal consent from their families will be filled with a personal information form, asthma control test and quality of life scale for children. The standard care and treatment of the asthmatic child included in the experimental group will be continued without any intervention. The child included in this group will be taught the Buteyko Breathing Technique (BST) via a smart phone, and the training video will be watched and taught. The training video will be watched on the official site that explains BST in a practical way. The video will be downloaded to the phone of the child or parent using a smartphone at home, for researchers to apply later at home. The participant will continue to apply this technique at home for 10 minutes in addition to his treatment when he needs a bronchodilator in the morning and evening for 4 weeks.
  Interventions: Behavioral: BUTEYKO RESPIRATORY TECHNIQUE
- GROUP WITH STANDARD CARE AND TREATMENT (No Intervention): This group consists of children aged 7-12 years with asthma who continue to receive standard care and treatment. Children with written and verbal consent from their families will be filled with a personal information form, asthma control test and quality of life scale for children. Asthma control test and quality of life scale for the child with asthma will be administered to the participant who continues the standard treatment and care for 4 weeks. After the research data are collected, the children in the control group will be shown a video explaining the BST in a practical way.

INTERVENTIONS:
Behavioral: BUTEYKO RESPIRATORY TECHNIQUE — Buteyko Breathing Technique In recent years, breathing exercises have been used as one of the non-pharmacological, alternative and/or complementary approaches in the management of many chronic diseases and conditions. Buteyko Breathing Technique (BST), Russian Dr. It was developed by Konstantin Buteyko in the 1950s. Dr. Buteyko evaluates the normal respiration over carbon dioxide, the respiratory holding time used in the technique is defined as a control pause, and this value shows the body's oxygenation and carbon dioxide tolerance. BST is a technique performed only through the nose, which includes respiratory control and respiratory hold after inhalation.
  Arms: BUTEYKO RESPIRATORY TECHNIQUE APPLIED GROUP

SUMMARY:
In this study, the effect of buteyko breathing technique applied in children aged 7-12 years with asthma disease on asthma control and quality of life is examined.

Asthma is a serious global health problem affecting all age groups. In studies conducted with the ISSAC (International study of asthma and allergies in childhood) method, the prevalence of asthma varies between 4-23% in developed populations. In childhood prevalence studies in our country, the cumulative asthma prevalence was found to be between 13.7% and 15.3%.

There are personal and environmental factors of genetic origin that cause asthma. Its prevalence is increasing in many countries, particularly among children. Asthma is a chronic inflammatory disease of the airways in which many cells and cellular elements play a role. It is seen with recurrent episodes of wheezing, coughing and shortness of breath due to lower airway obstruction and chronic inflammation.

Nurses will contribute to the protection and improvement of patients' health and well-being, to control asthma, to increase the quality of life, and to reduce health care expenditures, thanks to the hands-on training they will give to patients with asthma.

Keyword: Asthma, Quality of Life, Asthma Control

DETAILED DESCRIPTION:
Asthma; It is a chronic disease characterized by wheezing, shortness of breath, and cough symptoms, resulting from airway inflammation, airway hyperresponsiveness, and varying degrees of airway obstruction.

Asthma is a serious global health problem affecting all age groups. Its prevalence is increasing in many countries, particularly among children. Asthma affects the society not only economically but also socially. It is an important cause of school and workforce loss all over the world.

According to the National Burden of Disease Studies, the burden of disease caused by asthma in our country is ninth in rural areas and 14th in urban areas. Studies suggest that deaths caused by asthma can be prevented.

Although there is no clear relationship between prevalence and mortality in studies on asthma in the world, approximately 300 million people in the world are affected by asthma. However, it is thought that asthma is the cause of one of every 250 deaths in the world. It is estimated that 250,000 people worldwide die from asthma in one year.

Childhood Asthma Childhood asthma is characterized by chronic airway inflammation. It is defined by a history of respiratory symptoms such as wheezing, shortness of breath, cough, and chest tightness, with variable expiratory airflow limitation.

Chronic inflammation of the airways is characterized by recurrent morning and night cough and chest tightness in children. These inflammations are explained by airway structural cells such as T lymphocytes, smooth muscle endothelial cells and eosinophils. Airway obstruction caused by asthma attack in children is controlled with drugs.

Asthma in Children and Nursing Management in Asthma Attacks Asthma, which is a chronic disease, also affects the social and family lives of children in the community. Due to the increasing symptoms over time, the child begins to have difficulty in performing social and daily activities. The frequency of treatments causes the child to go to school, communicate with friends, and reduce the time spent in games and entertainment. In the process of chronic diseases, problems are experienced due to the inability of parents to go to work and the increase in the financial burden of the family.

Symptoms of recurrent asthma attacks may cause difficulties in performing daily activities (movement, nutrition, excretion, hygiene, sleep, etc.), intensification of emotional stress, and increased dependence on others.

The aim of nursing care in asthma in children should be to increase their control over their diseases by providing acceptance of the disease and compliance with treatment. This will increase the children's self-confidence. For this, the nurse should remove the uncertainties about the disease and provide education about prevention and drug effects to reduce daily symptoms and attacks. In this context, nursing interventions should be based on preventing attacks and symptoms, supporting them to have normal lung function and their participation in home, work, school and exercise activities.

Buteyko Breathing Technique In recent years, breathing exercises have been used as one of the non-pharmacological, alternative and/or complementary approaches in the management of many chronic diseases and conditions. Buteyko Breathing Technique (BST), Russian Dr. It was developed by Konstantin Buteyko in the 1950s. Dr. Buteyko evaluates the normal respiration over carbon dioxide, the respiratory holding time used in the technique is defined as a control pause, and this value shows the body's oxygenation and carbon dioxide tolerance. BST is a technique performed only through the nose, which includes respiratory control and respiratory hold after inhalation. The main purpose of the technique is the controlled prolongation of respiration, including control pauses/respiratory hold periods for the purpose of extending this time over time.

Breathing exercises are widely used in lung diseases. Many positive results have been reported in studies. In these studies, it has been shown that in patients with moderate or severe asthma who received inspiratory muscle training, improvement in asthma symptoms, decrease in β2-agonist use, decrease in emergency department admissions and hospitalizations, and increase in recovery rates from the hospital.

By using the Buteyko method instead of bronchodilators, it is aimed that patients can control their symptoms (such as chest tightness, wheezing) and reduce the frequency and severity of symptoms. It has been reported that with the application of this method, asthmatic patients experience less mucus formation, less chest tightness, better sleep, feel more energetic, and use less medication.

İmportance The increase in access to treatment and options in the world and in Turkey causes a decrease in deaths due to the disease. However, with the increase in people's actions to stay healthy, the problem of combating chronic diseases comes to the fore.

Asthma is a serious global health problem affecting all age groups. There are personal and environmental factors of genetic origin that cause asthma. Its prevalence is increasing in many countries, particularly among children. National and international asthma guidelines have been prepared in order to optimally control the disease in patients with asthma.

In cases where asthma is not controlled, it negatively affects the physical, psychological and social lives of patients.

In children with asthma, it is necessary to determine the factors that cause attacks and initiate symptoms, to take measures to protect them and to follow up at regular intervals. As health personnel, nurses have important duties in this regard.

Contribution In the light of this information, the effect of the Buteyko Respiratory Technique, which has not been done much in Turkey yet, will be evaluated for the effect of asthma, which is a chronic disease. The effectiveness of the applied technique will be evaluated using the Children's Asthma Control Test (CISAT) and Children's Asthma Quality of Life Scale (ÇAYKO) scales.

ELIGIBILITY:
Inclusion Criteria:

* with asthma,
* 7-12 years old with asthma
* Those who were diagnosed with asthma at least 6 months ago were treated

Exclusion Criteria:

* No asthma,
* Those over 12 years old and under 7 years old with asthma
* Any disease that will prevent or prevent the practice of breathing technique

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test for Children (CISAT) | at the end of 4 weeks
  Asthma control test is the most used test today, is easily understood by patients and their families, and is an important test that shows whether asthma is good or bad. AKT is a questionnaire consisting of 5 questions.
  It is a 5-item asthma control questionnaire that defines children whose asthma is not adequately controlled. The ACT is scored on a scale of 1-5 for each question.
  Patients rate each question between one and five points. The total score of the five questions forms the test result. If the total score is 25, it is considered as full control, 24-20 as partial control, and ≤19 as not under control

SECONDARY OUTCOMES:
The Scale of Quality of Life in Children with Asthma ÇAYKÖ | at the end of 4 weeks
  ÇAYKÖ Juniper et al. It was developed by Yuksel et al. made by ÇAYKÖ consists of 3 sub-units and 23 questions: 'symptoms', 'activity limitation' and 'emotional function'. The 'symptoms' sub-unit consisting of 10 questions (4, 6, 8, 10, 12, 14, 16, 18, 20 and 23) questions shortness of breath, wheezing, cough, chest tightness, and fatigue. In the "emotional function" sub-unit consisting of 8 questions (5, 7, 9, 11, 13, 15, 17 and 21), emotions such as sadness, resentment, fear, anxiety, anger, feeling different or excluded are questioned. In the 'activity restriction' sub-unit (1, 2, 3, 19 and 22) consisting of 5 questions, physical, social, school and sleep statuses are questioned. At the beginning of the study, the patient was asked to choose the 3 most difficult activities out of 39 activities during the last week.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Balcali Hospital Adana, Adana
  - Çukurova Üniversitesi Balcalı Hastanesi, Adana

IPD SHARING:
Plan to Share IPD: No